CLINICAL TRIAL: NCT07085871
Title: A Randomized Controlled Trial to Assess the Impact of School Meals Including Fish Powder on the Nutritional Status and Diet Quality of Malawian Schoolchildren
Brief Title: Nourishing for Knowledge: Fish Powder in School Meals in Malawi
Acronym: FAO/LUANAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Agriculture Organization of the United Nations (FAO) (Other)
Collaborators: Institute of Marine Research (Other); University of Bergen (Other); Lilongwe University of Agriculture and Natural Resources (LUANAR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FAOFVCGLO188MUL; Project Code: FVC/GLO/188/MUL (Other: Food and Agriculture Organization of the United Nations)
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Zinc Concentration in DBS
Keywords: Fish; Fish powder; schoolchildren; zinc; DBS

STUDY DESIGN:
Intervention Model Description: The study has been planned as a two-armed single-blinded RCT with a closed cohort design, featuring two parallel groups with a 1:1 allocation ratio for intervention and control groups. The intervention group will receive the normal school meal with 3-5g of fish powder added to it, while the control group will receive the school meal as normal (with no added fish powder).
Who Masked: Participant, Care Provider
Masking Description: This RCT is single-blinded, thus students will remain blinded throughout the duration of the RCT, so as not to affect their normal behavior in relation to food consumption or the perception of some students receiving a "superior" meal than others. Unblinding will only be done in cases where it is necessary, for example, if adverse effects are recorded during monitoring and knowledge on which treatment the student receives is relevant.
  The research team will not be blinded, but access to personal data will be restricted to only grant access to data necessary for implementation. Compliance supervisors in the study schools will have access to the list of students enrolled in the study in the school where they are located, and the allocation of those students in the treatment and control group. The Trial Manager will have access to the full list of students enrolled in the study across all schools, and their allocation to treatment or control group. Researchers at the Institute of Ma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School Meal + Fish Powder (Experimental): The intervention meals will aim to align with the nutrition standards defined by the Government of Malawi, or those developed by FAO and WFP if none are available. Recipes have been developed in line with the Government of Malawi and WFP Home-Grown School Feeding Recipe Book. The total weight of the dried ingredients in the control and treatment meals is equal in the two scenarios proposed below (i.e. there is a direct substitution of ingredients - 5 g of groundnut flour is substituted for 5 g of fish powder in the treatment meals). This was done as school feeding programs are usually on a tight budget, and adding more food may not be feasible. Thus, the total amount of food is not changed, but the number of ingredients increases by one, to include fish powder.
  Interventions: Other: Fish Powder
- Normal School Meal (No Intervention): This arm will receive the school meal as normal, with no additional ingredient.

INTERVENTIONS:
Other: Fish Powder — This RCT aims to test the effectiveness of fish powder (produced from dried fish from Lake Malawi - Lake Malawi sardine) used to fortify school meals. The intervention meal will be the normal school meal, however substituing 3-5g of ingredients (such as soya flour, maize flour or groundnut flour) for 3-5g of fish powder.
  Arms: School Meal + Fish Powder

SUMMARY:
Background: This randomized controlled trial (RCT) is a research component of a Food and Agriculture Organization of the United Nations (FAO) project in Malawi. The project aims to initiate pilot programs to integrate fish powders into existing home-grown school feeding program frameworks and meals served in selected schools in Malawi. The objective of the RCT is to assess the impact on dietary diversity and nutrition status (through biomarker analysis) of children receiving school meals in selected pilot schools.

Trial Design: This will be a two-armed single-blinded RCT with a closed cohort design, featuring two parallel groups with a 1:1 allocation ratio. The intervention will include 3-5g of fish powder added to the school meal (per 100g serving) five days per week, while the control group will receive the usual school meal. Children (n=270) of at least 10 years of age will be enrolled in the study. The primary outcome variable is the difference between the two arms in the contribution of school meals to zinc concentration measured in dried blood spots (DBS).

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will be implemented as a research component of the Food and Agriculture Organization of the United Nations (FAO) Flexible Voluntary Contribution fund (FVC) Sub-program entitled "Strengthening Capacity of Small-Scale Aquatic Food Producers for School Food and Nutrition". Starting in 2025, the Sub-program aims to initiate pilot programs to integrate aquatic food products into existing home-grown school feeding program frameworks and meals served in selected schools. The Sub-program has a research component, which will include an RCT in one country (Malawi) to assess the effectiveness of, and monitor the inclusion of, aquatic food products (specifically, fish powder) in school meals in schools participating in the pilot program. The objective of the RCT is to assess the impact on dietary diversity and nutrition status of children receiving meals from schools participating in the pilot program.

This will be done through collection of dried blood spot (DBS) samples pre- and post-intervention, to determine changes in nutritional status using biomarkers for key nutrients which may be attributed to increased fish consumption. The inclusion of fish powder in school meals will be monitored for compliance with the study protocol. Additionally, questionnaires will be administered to assess dietary diversity of schoolchildren to understand changes in nutritional status in the context of the whole diet.

Samples of the fish powders and porridges served in pilot schools will be collected for food composition analysis. Analysis of food composition will be conducted in an accredited laboratory to determine nutrient content of the fish powder, as well as the control (regular school meal) and intervention meal (regular school meal with fish powder added). These data may be used to demonstrate linkages between nutritional composition of fish products / meals and changes in nutritional status of schoolchildren consuming fish powder in school feeding programs.

Supplementary data on the costs and benefits to fish processors supplying fish powder to schools will be collected under the FAO FVC Sub-program.

Implementation of the RCT will be managed by a Trial Manager to be recruited by LUANAR, and supervised by the Principal Investigator and Lead Researcher listed below:

* Principal Investigator (PI): Professor Alexander Kalimbira (Department of Human Nutrition and Health, LUANAR)
* Lead Researcher, FAO: Molly Ahern (Fisheries Officer from the Food and Agriculture Organization (FAO) Fisheries Division's Food Safety, Nutrition and Health team) The study will be done in collaboration with relevant local partners (Malawi Department of Fisheries, Ministry of Education, Ministry of Health, World Food Programme, Malawi Bureau of Standards), and with guidance from identified experts from other institutions, such as University of Bergen (Norway) and Institute of Marine Research (Norway). The CVs of the PI, Lead Researcher and experts from collaborating institutions are included as appendices to the protocol.

Problem Statement / Rationale and Justification Aquatic foods can contribute greatly to nutrition but are often lacking from diets of the most vulnerable. Micronutrient deficiencies are persistent in Sub-Saharan Africa, contributing to serious public health issues (Stevens et al. 2022). Aquatic foods are rich in multiple micronutrients such as vitamins A and B12, iron, and zinc and are one of few natural dietary sources of vitamin D3, iodine, and eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) (two long-chain polyunsaturated fatty acids), which are often lacking in the diets of vulnerable populations. The fatty acids unique to aquatic foods, together with iodine, are necessary for cognitive development, not only during the first 1000 days but also in particular times of adolescence (referred to as "brain spurts") (Thatcher, 1991).Based on FAO Food Balance Sheets, per capita consumption of aquatic foods in Malawi is 10.1kg per annum, less than half the global average (FAO, 2024). Micronutrient deficiencies persist even in countries with relatively high aquatic food consumption, thus pointing to questions relating to quality of the aquatic foods consumed, quality of dietary intake data, or dietary equality, as per capita figures are based on averages and do not consider distribution of foods within the country, community or even within a household. Studies have shown that children's diets in Malawi are sub-optimal, e.g. only nine percent of children aged 6-23 months met minimum acceptable diet (National Statistical Office (NSO) 2021), and very few consume animal source foods such as fish. This is often due to lack of knowledge on the importance of fish for nutrition, or how to incorporate fish into the diets of young children. Several studies have shown that powder made from dried fish can be easily added to existing local recipes, is nutrient-rich (Abbey et al., 2016; Byrd et al., 2021, Bogard et al., 2015), acceptable in diets of young children in many countries (Glover-Amengor et al., 2012), including Malawi (Ahern et al., 2020), and has extended storage life (Ngóng'ola-Manani et al., 2020).

School meal programs offer an entry point for nutrition programs and introducing healthy diets; however they often lack nutritious foods such as fish and other aquatic foods. HGSF programs source ingredients locally but lack foods such as fish, often citing issues such as food safety and cost (Ahern et al. 2021). While there is general recognition that fish and aquatic foods are beneficial for nutrition, the potential benefits of inclusion of aquatic foods in school meal programs (and particularly HGSF programs) have not been studied. HGSF programs offer an entry point for encouraging healthy diets for schoolchildren and community development and contribute to the realization of sustainable development goals (SDGs) 1, 2, 3, 5, 12 and 14. The importance of HGSF for poverty alleviation (SDG1) and zero hunger (SDG 2) have been recognized by the UN Hunger Task Force as well as regional bodies such as African Union Development Agency - New Partnership for African Development (AUDA-NEPAD 2020).

Consumption of animal-source food such as fish with plant-source foods can have an enhancing effect on micronutrient absorption, but questions remain on how small quantities of fish can result in this effect. Consumption of aquatic animal-source foods can improve micronutrient absorption (particularly iron and zinc) from plant-source foods when consumed together (Consalez et al., 2022). Although several publications (Kawarazuka 2010; Kawarazuka and Béné 2011; Byrd et al. 2022; Michaelsen et al. 2009) point to the potential nutritional benefit of small amounts of fish added to meals, there is no empirical evidence. Little is known about the impact on nutritional status made by consumption of low doses of aquatic foods. The minimum quantity of fish that (Consalez et al. 2022) found evidence of for the enhancement of micronutrient absorption from plant-source foods was 40g . This RCT has high ecological relevance due to its real-life setting, as the low dosage of fish powder included in the intervention meal has been designed considering food preferences of schoolchildren, availability and accessibility of fish, and cost considerations for school feeding programs. The RCT will contribute to knowledge by exploring the dose-response relationship for low-dosages of fish (in powdered form) consumed regularly in school meals in selected regions and schools in Malawi .

There is need for evidence of the impact of school meals on nutrition status of schoolchildren, as well as nutrient content of locally produced foods in comparison to imported foods served in schools. The Global Child Nutrition Foundation (GCNF) survey of school meal programs in Malawi defined two key research priorities, including assessing students' nutritional status and class performance and investigating the difference in availability and nutrient content between locally produced foods and imported foods used in school feeding programs (GCNF 2018). Furthermore, there is a lack of knowledge on dietary diversity of schoolchildren, and consumption of aquatic foods in this critical period of growth, particularly through school feeding programmes. This RCT aims to fill these gaps, to build evidence of the nutritional importance of aquatic foods in school meals and contribute to knowledge on diets of schoolchildren in Malawi. The nutrient content of school meals served during the RCT will also be analyzed, contributing to knowledge on nutrient content of locally produced and imported foods used in school feeding programs.

In the past, insufficient funding has resulted in an inability to gather strong evidence of the importance of aquatic foods in school meals in LICs. Pilot programs including aquatic foods in school meals have been implemented by FAO and others in the past through small projects with limited funds, however little is known about the costs and benefits of these programs for consumers and producers. This lack of scientific evidence on costs and benefits to consumers and producers impacts sustainability of these initiatives beyond the termination of project funding. This RCT will complement the FAO FVC Sub-program by contributing to evidence on the costs and benefits of locally produced fish powder used in school feeding pilot programs in Malawi, to provide information which may support decision-making regarding longer-term sustainability of HGSF programs including aquatic food products (see Objectives and Methodology for further information).

Study Objectives The aim of the study is to assess the effects of school meals fortified with locally-produced fish powder on diet quality and nutritional outcomes of schoolchildren in selected Malawian schools, as compared to conventional school meals served in HGSF.

* Objective 1: Measure changes in zinc status of schoolchildren enrolled in a two-armed RCT
* Objective 2: Measure changes in micronutrient status of schoolchildren enrolled in a two-armed RCT
* Objective 3: Using questionnaires, assess changes in dietary diversity of schoolchildren

Methods / Experimental Design RCT Design The study has been planned as a two-armed single-blinded RCT with a closed cohort design, featuring two parallel groups with a 1:1 allocation ratio for intervention and control groups. The intervention group will receive the normal school meal with 3-5g of fish powder added to it, while the control group will receive the school meal as normal (with no added fish powder).

Null Hypothesis: Fish powder addition to school meals does not change zinc concentration measured in DBS collected from schoolchildren.

Alternative Hypothesis: Fish powder addition to school meals changes zinc concentration measured in DBS collected from schoolchildren.

Intervention and Study Period The intervention will take place during the 2026 school year, likely in the third school term, which runs from May to July. The timing was considered appropriate, as it is a time of year where fish are highly available from Lake Malawi and coincides with one school term. In the case that the intervention cannot take place in this school term, it will be conducted in the following school term, between September and December 2026. The overall FAO FVC Sub-program aims to work with fish processors to process fish powder at times of high fish availability and package and store fish powder so that sufficient quantities are available for the duration of the study.

Schools will receive grant money to purchase fish powder to be added to existing recipes used in schools, and school staff will be trained to prepare recipes. Fish powder was identified in a formative study completed by FAO and LUANAR (2023) as an acceptable product both for schoolchildren who participated in an acceptability trial as well as school health and nutrition staff, who noted its ease-of-use with existing school meal program recipes. These results are published (Ahern et al., 2025). The Sub-program in which this RCT is nested will work with small-scale fish processing organizations in target districts to build capacity to supply safe fish powder to identified intervention schools. Prior to the start of the study, microbial and chemical analyses of the fish powder will be conducted to ensure that they are safe to consume, based on maximum allowable limits determined by the Malawi Bureau of Standards (MBS). Additionally, samples of the fish powder and control and treatment porridges will be collected for nutrient analysis. High-quality analytical data on the food composition of the cooked porridges is very valuable to this study, as it will provide information on the nutrients actually reaching the schoolchildren and will aid in interpreting the biomarker analysis.

The aims of this study align well with the Government of Malawi's School Health and Nutrition Guidelines (Ministry of Education Science and Technology, Ministry of Health, and Ministry of Agriculture and Food Security 2009) which emphasize the importance of locally acceptable and locally sourced foods that can be easily and quickly prepared for large numbers of learners. The intervention meals will aim to align with the nutrition standards defined by the Government of Malawi, or those developed by FAO and WFP if none are available. The total weight of the dried ingredients in the control and treatment meals will be equal (i.e. there will be a direct substitution of ingredients - for example, 5 g of groundnut flour is substituted for 5 g of fish powder in the intervention meals). This is proposed as school feeding programs are usually on a tight budget, and adding more food may not be feasible. Thus, the total amount of food is not changed, but the number of ingredients increases by one, to include fish powder.

Implementation in Schools The meals will follow the existing meal schedule, as they will be provided once a day at breakfast time 5 times per week for all the schoolchildren independent if they are part of the 270 students that will take part in the RCT. All schoolchildren will receive their regularly scheduled school meal, while data (DBS samples and dietary recall data) will only be collected from the 270 students who are enrolled in the RCT. The RCT will be conducted for a total of one school term, or three months (or 12 weeks). The intervention will include 3-5 g of fish powder (per student) added to school meals (to be based on quantity of cereals served, not to exceed 5% fish powder by total weight of cereal + fish powder ), while the control group will receive meals as normal. Two large pots will be used to cook the morning porridge, one including the intervention meal (regular school meal with fish powder added) and one with the control meal (regular school meal). Enrolled study participants will be blinded as to which meal they will receive. Large pots are used to prepare the porridge each morning by volunteers from the community. Each pot serves approximately 400 portions of porridge. Thus, depending on enrolment numbers, at least 2 pots of porridge will be made per school each day. One pot of porridge will be the usual school meal (or control) and the other pot will include the fish powder added to the usual meal (or intervention). Reusable plastic plates will be purchased in two colors, with children assigned to the intervention group receiving one color of plate (for example, red) and the children in the control group receiving the second color of plate (for example, blue). Children not enrolled in the study can choose either colored plate (except for those with known allergies to fish, see below). To ensure compliance, 1 member of the research team (from here on, referred to as the compliance supervisor) per school will be present at mealtime every day to ensure that students assigned to the control and intervention groups have the correct colored plate and receive the correct meal (control or intervention). Further information on monitoring for compliance is detailed in the section on Compliance Monitoring.

The school meals including fish powder will be prepared by school cooks, usually women members of the community, that are already involved in preparation of school meals. They will receive at least two training sessions to ensure that meals are prepared according to the menus and recipes developed. A package of materials has been developed for the trainings based on the results of a capacity needs assessment carried out under the FAO FVC Sub-program, which identified key capacity gaps at school level for providing nutritious meals to students.

To support implementation and acceptability of the school meals with fish powder added, a series of simple educational activities, focusing on the nutritional importance of fish and aquatic foods will be implemented in the intervention schools, targeting children of at least 10 years of age.

The strategy has been designed following FAO's model for school-based food and nutrition education (FAO 2020), as well as the Malawi Government's School Health and Nutrition Guidelines (Ministry of Education Science and Technology, Ministry of Health, and Ministry of Agriculture and Food Security 2009), which emphasize the importance of integrating nutrition education into curriculum and activities to help learners, teachers and communities to choose a wide variety of foods as part of their diets.

Sample Size The mean (64.85 µg/dL) and standard deviation (±34.71) of zinc concentration (measured in serum) of school-aged children (5-14 years) was obtained from the Malawi Micronutrient Survey (2015/16) 'Other Biomarkers' dataset available through the DHS data portal. An effect size of 0.20 (corresponding to approximately 13 µg/dL) can be detected with a power of 80% and a significance level of alpha = 0.05 by studying 112 students per group (total n= 224) with 1:1 allocation. Calculations were made using clincalc.com RCT sample size calculator, considering two independent study groups and a continuous primary endpoint. A total of 270 students will be enrolled in the study, to account for a 20% dropout rate.

Randomization Sequence Generation Participants will be randomly assigned to either control or experimental group with a 1:1 allocation as per an excel-generated randomization stratified by site (school).

Allocation Concealment mechanism The trial manager will be responsible for recruiting 270 students to participate in the study. Once recruited, the trial manager will record the name, age at baseline and the location (school) of the student in an Excel file. This file will be shared with FAO to assign ID numbers for each student, including a letter for their school and a number for the individual (for example, A01, B12, etc.) The ID numbers will be copied into another Excel file and given a corresponding random number (0-1) generated by the Excel function Rand(). The ID numbers will be sorted by the random number in ascending order, and the first half of ID numbers for each school will be allocated to the treatment group, while the second half will be allocated to the control group.

Implementation A blinded member of the research team (at FAO / University of Bergen) will generate the independent allocation sequences and randomization lists for each school. The Trial Manager (at LUANAR) will be responsible for enrolment of students in the study and will have access to the lists of students in each treatment group, stratified by school, in order to implement the trial and ensure compliance. Compliance supervisors in the study schools will have access to the list of students enrolled in the study in the school where they are located, and the allocation of those students in the treatment and control group, to ensure compliance to the allocated meal.

Blinding This RCT is single-blinded, thus students will remain blinded throughout the duration of the RCT, so as not to affect their normal behavior in relation to food consumption or the perception of some students receiving a "superior" meal than others. Unblinding will only be done in cases where it is necessary, for example, if adverse effects are recorded during monitoring and knowledge on which treatment the student receives is relevant.

The research team will not be blinded, but access to personal data will be restricted to only grant access to data necessary for implementation. Compliance supervisors in the study schools will have access to the list of students enrolled in the study in the school where they are located, and the allocation of those students in the treatment and control group. The Trial Manager will have access to the full list of students enrolled in the study across all schools, and their allocation to treatment or control group. Researchers at the Institute of Marine Research will have access to the analyzed biomarker data, which will be identified using ID numbers. Only the lead researcher at FAO will have access to both the list of students with ID numbers, assigned allocation groups and the analyzed biomarker data, for purposes of assessing outcomes.

Statistical Methods A simple t-test will be used to analyse the significance of the results between the two arms of the RCT for the primary outcome variable of zinc concentration. Any potential bias should be accounted for in the randomization, thus further analysis should not be necessary.

Data Collection In addition to measurements of zinc concentration and other key nutrients (using biological samples - dried blood spots), a questionnaire will be used to collect data on the background diets of children and some demographic information. The protocol for biological sample collection, as well as the questionnaire for children enrolled in the study are included as appendices to this study protocol.

Dietary and sociodemographic data of the study participants will be collected pre-intervention (before the start of the school term) and will be repeated after the RCT is completed, at the end of the school term (post-intervention). Schoolchildren of at least 10 years of age will complete a structured questionnaire on household sociodemographic characteristics, administered by trained enumerators. The child's caregiver may be present for the data collection, but the questionnaires are designed so that a child of at least 10 years of age may answer all of the questions on their own.

The dietary assessment will involve three methods: a list-based 24-hour dietary recall to assess children's total diet, a food frequency questionnaire for each food group, and a semi-quantitative recall of fish consumption. The 24-hour diet recall method requires children to recall all foods and beverages, except water, consumed on the previous day from when they woke up to when they went to sleep. This is a quick recall of all foods eaten during the previous day generated by the child, and will be assisted using the list-based method, using food lists developed for Malawi (for example, asking the child, "Yesterday, from the time you woke up to the time that you went to sleep at night, did you consume any cereals, roots or tubers, such as mpunga (rice), vingoma (maize), etc… ).

If necessary, the dietary recall may be aided by the child's main caregiver (if the caregiver / guardian may be present during data collection). Interviewers will then probe for more complete information about foods recorded on the quick list by asking questions like- "Do you remember eating or drinking anything else?", and "Did you add anything else to this food?" This approach will gather more detailed information on each food item consumed including portion sizes (with the aid of food models and handy household measures), recipes, and final review and double-check for potentially missed foods. The place of consumption will focus on household consumption, as food consumption in school will be tracked separately by Compliance Supervisors who are part of the research team. The dietary recall interviews will be conducted by trained local field assistants knowledgeable about foods available in the marketplace and about local preparation practices. The field assistants will use validated food models and handy measures / visual aids to facilitate the recall process.

The visits for the data collection will be scheduled from Tuesday to Saturday to capture the school weekdays (Monday-Friday).

Data Management Treatment Allocation and Personal Data Researchers, students and supervisors who have access to personal data have a duty of confidentiality, thus procedures for processing personal data will be followed. These procedures include de-identifying personal information such as names, birth dates and other personal identifiers by replacing them with a number or code, and / or anonymizing data by removing names, birth dates or other unique characteristics.

Access to personal data for members of the research team will be restricted, granting access for different members of the research team only to data considered necessary for implementation. Compliance supervisors in the study schools will have access to the list of students enrolled in the study in the school where they are located, and the allocation of those students in the treatment and control group. The Trial Manager will have access to the full list of students enrolled in the study across all schools, and their allocation to treatment or control group. Researchers at the Institute of Marine Research will have access to the analyzed biomarker data, which will be identified using ID numbers (no personal data). Only the lead researcher at FAO will have access to both the list of students with ID numbers, assigned allocation groups and the analyzed biomarker data, for purposes of assessing outcomes.

All data will be stored electronically in an encrypted folder that is accessible through an encryption key which will be made available to the lead researchers from FAO, LUANAR and IMR / University of Bergen named in the protocol submitted and approved by the LUANAR Research Ethics Committee. Personal data will not be stored longer than what is necessary to carry out the RCT. De-identified or anonymized data may be stored by the FAO beyond the RCT, following terms of privacy regulations.

Data collected in Questionnaires for Schoolchildren and Monitoring of School Meals The questionnaire for schoolchildren and the questionnaire for monitoring school meals (available as appendices to this study protocol) will be uploaded into Kobo Collect, an application for computer-assisted personal interviews (CAPI), to facilitate data collection and data entry. Kobo Collect can be downloaded on any Android device and allows data collection even while the device is online. Data will be uploaded to the Kobo server each day to allow the Trial Manager and research team to monitor compliance across schools. Access to the data uploaded to the Kobo server will be restricted to the limited members of the research team.

Data Analysis and Dissemination of Information Pre-intervention samples of DBS will be sent to the selected Laboratory and stored until post-intervention samples of DBS are also received. Analysis of pre- and post-intervention samples will take place at the same time, to ensure that they are completed under the same conditions. The results of DBS analysis, as well as dietary recall data and compliance monitoring data will be analysed by FAO, in collaboration with LUANAR and collaborating institutions (University of Bergen and Institute of Marine Research Norway).

Dietary recall data will be analysed by calculating individual dietary diversity scores based on (FAO 2021). Data collected on compliance will be analyzed to provide key indicators, such as average portion size served per student, and percentage of meal consumed.

Results will be communicated back to communities and national stakeholders, as well as in international conferences where relevant, and synthesized in scholarly journal articles.

Ethical Considerations The trial will be conducted in accordance with the declaration of Helsinki and will be registered in Clinical Trials. The study will be a parallel group, two-arm single-blinded RCT. Ethical considerations were considered, such as that of providing different meals to different students within the same school which includes potential singling out of pupils and providing meals that could be perceived as 'better' to only a few students. To address these ethical concerns, blinding of students participating in the study will be done, with only the compliance supervisor at the study site and the research team outside of the study site knowing which students receive the intervention or control meal. The compliance supervisor present in the study site will monitor mealtime to ensure compliance of enrolled participants to allocated groups, as well as other information as detailed in the study protocol (negative reactions, etc.) Inclusion Criteria While all students in the school will be served a school meal (either control or intervention meal), only students of at least 10 years of age will be enrolled in the study. This age limit for inclusion is based on two criteria; first, due to logistical reasons, as the data collection will likely take place at the school, where the caregiver / guardian of the child may not be able to be present. Consent will be sought from the child's guardian prior to enrolment in the study, as well as assent from the child. Secondly, the age limit of at least 10 years of age is based on studies showing that this is the minimum age that children can recall their diet accurately.

Informed Consent and Awareness Raising As the RCT involves processing of personal data, ethical clearance was obtained from the LUANAR Research Ethics Council. Additionally, awareness raising of the study will be conducted amongst caregivers of children at the school, and informed consent will be sought for each student enrolled in the trial from the child's caregiver. The consent must be informed, voluntary and documented, and may be withdrawn at any time during the execution of the RCT. Consent forms will be provided on paper, in the local language, and signed consent forms will be scanned and stored. In addition, the children will also be asked to assent to the study. Assent will be informed, voluntary, and documented, and may be withdrawn at any time during the execution of the RCT. Any child with allergies to fish products will be excluded from the study and will receive the same-coloured plate as the control group to ensure that they are not served the meal with fish powder added.

Benefits, Risks and Risk Management The benefits of the treatment meal in comparison to the control meal are unknown, as the difference between treatment and control meals will be the substitution of a very small quantity of groundnut flour for fish powder. While consumption of fish is generally understood to be beneficial, there are no known experimental studies that have evidenced benefits from consumption of small amounts of fish.

To mitigate risks relating to food safety, the fish powders will be analysed to ensure food safety prior to the trial starting. To ensure quality of fish powders, the FAO project aims to work with fish processors to develop standard operating procedures which follow Good Hygiene and Good Manufacturing Principles (GHP and GHP) in fish value chains.

ELIGIBILITY:
The selection of study sites in Malawi will be delimited by two criteria. Firstly, the schools have to be currently implementing a full home-grown feeding modality, where food and ingredients are purchased directly by schools using government, Mary's Meals or WFP funds, given that this modality has been endorsed by the Government of Malawi. All schools that do not implement school meals, are privately funded or implement meals with hybrid or traditional school feeding modalities will be therefore excluded.

Secondly, as HGSF programs often require that foods are sourced within a given radius of the school, study sites will be limited to those where fish processing organizations are known to be present. Of these, three districts were selected (Mangochi, Salima and Karonga). As these three districts are lakefront districts, it was recognized that fish may be a more typical part of the diet of people in these districts than in upland districts (Simmance et al. 2022). Thus, one upland district (Dowa), further away from where known fish processing organizations are present, was also selected for testing the intervention.

A list of schools will be compiled with data on geographical location, total enrolment, school feeding modality and implementing entity for the four identified districts. For the students to be eligible to participate in the study, they have to be at least 10 years old, considering the minimum age that children can report on their own food consumption . No maximum age is included, as it may be expected that the majority of children enrolled are aged 10-14 years, however, older students who may still be in primary school will not be excluded. Due to the closed cohort design and the duration of the intervention of one term, no loss of students due to termination of the school cycle is expected. Students will be excluded if they have grave intolerances or food allergies or with health conditions that may affect their food consumption. All eligible children in this age group from the selected schools will constitute the sampling frame at the child level. Screening of students for eligibility will be led by the Trial Manager, to be recruited by LUANAR

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Zinc concentration in Dried Blood Spots | 3-4 month school term (as defined by Malawi school calendar)
  Difference between the two arms in the contribution of school meals to zinc concentration (mcg/dL) in DBS collected from selected school children.

SECONDARY OUTCOMES:
Micronutrient Status of children | 3-4 month school term (as defined by Malawi school calendar)
  Difference between the two arms in the contribution of school meals to micronutrient status of school children. The impact of the intervention on micronutrient status of schoolchildren will be tested using DBS. This aligns with targets set by the Government of Malawi in their nutrition guidelines for school meals (2009), which aim to reduce vitamin A deficiency and anaemia in school age children and maintain median urinary iodine levels in school children (100 mcg/L) (Government of Malawi, 2010).
Diet Scores | 3-4 month school term (as defined by Malawi school calendar)
  Differences in between the two arms in diet scores at end of intervention period using dietary diversity scores based on semi-quantitative, list based 24-hour recall and food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kalimbira, PhD, Principal Investigator — Lilongwe University of Agriculture and Natural Resources
Locations (3):
- Malawi (3):
  - School to be randomly selected prior to RCT, Mangochi
  - School to be randomly selected prior to RCT, Nkhotakota
  - School to be randomly selected prior to RCT, Salima

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to FAO project webpage. The RCT will be conducted as part of this project. — https://www.fao.org/in-action/fish-aquatic-food-school-meals/en